CLINICAL TRIAL: NCT04528355
Title: A Prospective Outcomes Study of Pediatric and Adult Patients With Non-Malignant Disorders Undergoing Umbilical Cord Blood, Bone Marrow, or Peripheral Blood Stem Cell Transplantation With a Reduced-Intensity Conditioning Regimen (PRO-RIC)
Brief Title: Data Collection Study of Patients With Non-Malignant Disorders Undergoing UCBT, BMT or PBSCT With RIC
Acronym: PRO-RIC
Status: Recruiting | Type: Observational
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, BMT-CT at CHP of UPMC and Professor of Pediatrics and Immunology, University of Pittsburgh, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY20070105
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Primary Immunodeficiency (PID); Congenital Bone Marrow Failure Syndromes; Inherited Metabolic Disorders (IMD); Hereditary Anemias; Inflammatory Conditions
Keywords: Severe Combined Immune Deficiency (SCID) with NK cell activity; Omenn Syndrome; Bare Lymphocyte Syndrome (BLS); Combined Immune Deficiency (CID) syndromes; Wiskott-Aldrich Syndrome; Leukocyte adhesion deficiency; Chronic granulomatous disease (CGD); Hyper IgM (XHIM) syndrome; IPEX syndrome; Chediak-Higashi Syndrome; Autoimmune Lymphoproliferative Syndrome (ALPS); Hemophagocytic Lymphohistiocytosis (HLH) syndromes; Lymphocyte Signaling defects; Congenital Amegakaryocytic Thrombocytopenia (CAMT); Osteopetrosis; Hurler syndrome (MPS I); Hurler syndrome (MPS II); Krabbe Disease, also known as Globoid Cell Leukodystrophy; Metachromatic leukodystrophy (MLD); X-linked adrenoleukodystrophy (ALD); Alpha Mannosidosis; Gaucher Disease; Thalassemia major; Sickle cell disease (SCD); Diamond Blackfan Anemia (DBA); Crohn's Disease; Inflammatory Bowel Disease; IPEX or IPEX-like Syndromes; Rheumatoid Arthritis
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Congenital Bone Marrow Failure Syndromes; Severe Combined Immunodeficiency; Syndrome; Wiskott-Aldrich Syndrome; Leukocyte adhesion deficiency type 1; Granulomatous Disease, Chronic; Hyper-IgM Immunodeficiency Syndrome; Immune Dysregulation, Polyendocrinopathy, Enteropathy, X-Linked Syndrome; Chediak-Higashi Syndrome; Autoimmune Lymphoproliferative Syndrome; Lymphohistiocytosis, Hemophagocytic; Congenital amegakaryocytic thrombocytopenia; Osteopetrosis; Mucopolysaccharidosis I; Sudden Infant Death; Leukodystrophy, Globoid Cell; Leukodystrophy, Metachromatic; Adrenoleukodystrophy; alpha-Mannosidosis; Gaucher Disease; beta-Thalassemia; Anemia, Sickle Cell; Anemia, Diamond-Blackfan; Crohn Disease; Inflammatory Bowel Diseases; Arthritis, Rheumatoid | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: data collection — Study subjects will receive alemtuzumab, melphalan, thiotepa, fludarabine and hydroxyurea-based, reduced-intensity conditioning regimen in accordance with clinical practice at UPMC Children's Hospital of Pittsburgh at the discretion of the treating physician. Medical data will be abstracted from subject's medical charts once the patient signs the informed consent.

SUMMARY:
This is a data collection study that will examine the general diagnostic and treatment data associated with the reduced-intensity chemotherapy-based regimen paired with simple alemtuzumab dosing strata designed to prevented graft failure and to aid in immune reconstitution following hematopoietic stem cell transplantation.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) from a healthy donor can cure or alleviate a broad spectrum of non-malignant disorders (NMD). Although reduced-intensity conditioning (RIC) regimens promise decreased treatment-related morbidity and mortality, graft failure and infections are limiting the use of RIC in chemotherapy-naive patients. Dr. Szabolcs have completed several trials to evaluate a novel RIC regimen of alemtuzumab, hydroxyurea, fludarabine, melphalan, and thiotepa. The last trial at UPMC Children's Hospital of Pittsburgh of a highly effective and biologically rational chemotherapy-based RIC regimen paired with simple alemtuzumab dosing strata was tested and resulted in outstanding survival and remarkably low rates of graft failure. The favorable outcome described may serve as a toxicity and efficacy reference for emerging gene therapy strategies as well.

This prospective collection of clinical data will allow the investigators to further assess engraftment, GVHD, immunosuppressant use and overall survival in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patient, parent, or legal guardian must have given written informed consent.
2. Patient must be 2 months to 60 years (inclusive) of age at time of consent for all diagnoses.
3. Patients should have a non-malignant disorder amenable to treatment by stem cell transplantation, including but not limited to the following:

   A. Primary Immunodeficiency Syndromes
   * Severe Combined Immune Deficiency (SCID) with NK cell activity
   * Omenn Syndrome
   * Bare Lymphocyte Syndrome (BLS)
   * Combined Immune Deficiency (CID) syndromes
   * Combined Variable Immune Deficiency (CVID) syndrome
   * Wiskott-Aldrich Syndrome
   * Leukocyte adhesion deficiency
   * Chronic granulomatous disease (CGD)
   * Hyper IgM (XHIM) syndrome
   * IPEX syndrome
   * Chediak-Higashi Syndrome
   * Autoimmune Lymphoproliferative Syndrome (ALPS)
   * Hemophagocytic Lymphohistiocytosis (HLH) syndromes
   * Lymphocyte Signaling defects

   B. Congenital Bone Marrow Failure Syndromes
   * Congenital Amegakaryocytic Thrombocytopenia (CAMT)
   * Osteopetrosis

   C. Inherited Metabolic Disorders (IMD)
   * Mucopolysaccharidoses

     * Hurler syndrome (MPS I)
     * Hunter syndrome (MPS II)
   * Leukodystrophies

     * Krabbe Disease, also known as globoid cell leukodystrophy
     * Metachromatic leukodystrophy (MLD)
     * X-linked adrenoleukodystrophy (ALD)
   * Other inherited metabolic disorders

     * Alpha Mannosidosis
     * Gaucher Disease
     * Other inheritable metabolic diseases where HSCT may be beneficial

   D. Hereditary Anemias
   * Thalassemia major
   * Sickle cell disease (SCD)
   * Diamond Blackfan Anemia (DBA)

   E. Inflammatory Conditions
   * Crohn's Disease or Inflammatory Bowel Disease
   * IPEX or IPEX-like Syndromes
   * Rheumatoid Arthritis
   * Other inflammatory conditions where HSCT may be beneficial
4. Subjects receive either umbilical cord blood, bone marrow, or peripheral blood stem cell transplant with an alemtuzumab, melphalan, thiotepa, fludarabine and hydroxyurea-based, reduced-intensity conditioning regimen, according to clinical practice at UPMC Children's Hospital of Pittsburgh.

There are no exclusion criteria.

Ages: 2 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with Non-Malignant Disorders Undergoing Umbilical Cord Blood, Bone Marrow, or Peripheral Blood Stem Cell Transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of acute graft versus host disease (GVHD) | up to 5 years
  grades 3-4, chronic extensive GVHD
overall survival after HSCT | up to 5 years
  review of the existing medical records to check on the participant's survival status

SECONDARY OUTCOMES:
Describe degree of engraftment, based upon chimerism data | up to 5 years
  review of chimerism test results in the existing medical records to check on degree of donor engraftment measured by the percentage of donor-derived blood cells in the HSCT recipient
Describe probability to discontinue systemic immunosuppression medications | by 6, 9, and 12 months post-HSCT
  review of the existing medical records to check on the participant's current medications
Describe the tempo of immune reconstitution | over the first year post transplant
  review of the various test results in existing medical records to check on the participant's immune system recovery rate
Describe the use of donor leukocyte infusion (DLI) | up to 5 years
  review of the existing medical records to check on the participant's need for DLI

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — UPMC Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No